CLINICAL TRIAL: NCT01178892
Title: MsFLASH-02: Interventions for Relief of Menopausal Symptoms: A 3-by-2 Factorial Design Examining Yoga, Exercise, and Omega-3 Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Research on Women's Health (ORWH) (NIH); Nordic Naturals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MsFLASH-02; 1U01AG032699-01 (NIH); 1U01AG032682-01 (NIH); 3U01AG032699-01S1 (NIH); 1U01AG032669-01 (NIH); IR 7265 (Other: FHCRC IRB)
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hot Flashes; Menopause; Vasomotor Symptoms
Keywords: Hot Flashes; Menopause; Vasomotor symptoms; Yoga; Exercise; Omega-3; Fish oil
MeSH Terms: conditions — Hot Flashes; Motor Activity | interventions — Docosahexaenoic Acids; Yoga; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo; Behavioral: Yoga; Behavioral: Exercise; Behavioral: Usual Activity
- Omega-3 (Experimental)
  Interventions: Dietary Supplement: Omega-3; Behavioral: Yoga; Behavioral: Exercise; Behavioral: Usual Activity
- Yoga (Experimental)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Omega-3; Behavioral: Yoga
- Exercise (Experimental)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Omega-3; Behavioral: Exercise
- Usual Activity 1 (Other): Usual Activity 1 and Usual Activity 2 arms will be compared to the Yoga and Exercise arms.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Omega-3; Behavioral: Usual Activity
- Usual Activity 2 (Other): Usual Activity 1 and Usual Activity 2 arms will be compared to the Yoga and Exercise arms.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Omega-3; Behavioral: Usual Activity

INTERVENTIONS:
Dietary Supplement: Placebo — Three placebo gel capsules filled with vegetable oil are taken daily for a total of approximately 2 grams of vegetable oil. Each gel capsule also contains 15 IU of vitamin E, natural lemon flavoring, rosemary extract, and a small amount of non-omega-3 fish oil.
  Arms: Exercise; Placebo; Usual Activity 1; Usual Activity 2; Yoga
Dietary Supplement: Omega-3 — The study supplement, omega-3-fish oils, is taken as 3 gel capsules daily that together contain approximately 2 grams of fish oil. Each gel capsule (1/3 of the daily dose) has a total omega-3 dosage of 615 mg with two major omega-3 components of ethyl eicosapentaenoic acid (EPA; 425 mg) and docosahexaenoic acid (DHA; 100 mg). Vitamin E (15 IU), an antioxidant, is added to each gel capsule to prevent oxidation and preserve freshness. Each gel capsule also contains natural lemon oil and rosemary extract to enhance taste and freshness.
  Arms: Exercise; Omega-3; Usual Activity 1; Usual Activity 2; Yoga
Behavioral: Yoga — Yoga instruction is provided during 12 weekly 90-minute classes, designed for women without prior yoga experience. Each class includes an introductory breathing exercise, 11 to 13 gentle postures followed by deep relaxation with a visualization exercise. Study participants are expected to attend each of the 12 weekly yoga classes plus do daily 20-minute at-home practices. Classes are offered at 2 different times during the week.
  Arms: Omega-3; Placebo; Yoga
Behavioral: Exercise — The exercise intervention is facility-based aerobic exercise training on a treadmill, stationary bicycle or elliptical trainer performed 3 times a week for 12 weeks. The duration of each training session is determined for each woman based on the weekly total energy expenditure goal and workload required to achieve her prescribed exercise heart rate. Women train at 50-60% heart rate reserve (HRR) for the first month and then increase intensity to 60-70% HRR. To ensure that women train at their prescribed exercise heart rates, women wear Polar Heart Rate Monitors while exercising. The exercise counselor overseeing each exercise session records each participant's exercise heart rate every 5-10 minutes to document that she is in her target heart rate range.
  Arms: Exercise; Omega-3; Placebo
Behavioral: Usual Activity — Women randomly assigned to the "Usual Activity" group will be asked to continue with their usual physical activities during the study and not make changes. At completion of the intervention, women will have the opportunity to attend a yoga class and receive the yoga booklet, CD, and DVD for home use; or receive a one-month gym membership.
  Arms: Omega-3; Placebo; Usual Activity 1; Usual Activity 2

SUMMARY:
This study is the second clinical trial to be conducted by the Menopause Strategies - Finding Lasting Answers for Symptoms and Health (MsFLASH) research network, a group of investigators conducting clinical trials designed to find new ways to alleviate the most common, bothersome symptoms of the menopausal transition.

In this twelve-week clinical trial, 374 women aged 40-62 who are in the late menopausal transition or postmenopausal and experiencing bothersome hot flashes will be randomized to one of three behavioral intervention groups: yoga, exercise, or usual activity. All women will simultaneously be randomized to receive omega-3 supplementation or a matching placebo.

The primary aims of this trial are to compare the magnitude of changes in perceived, self-reported frequency and bother of vasomotor symptoms (VMS) before and after the intervention between yoga and the usual activity comparison group, between exercise and the usual activity comparison group, and between omega-3 fatty acid supplementation or placebo. The hypotheses to be tested are:

1. Women assigned to yoga will report lower frequency and less VMS bother than women assigned to the usual activity group at the end of a 12-week study period.
2. Women assigned to aerobic exercise at moderate-vigorous intensity will report lower frequency and less VMS bother than women assigned to the usual activity group at the end of a 12-week study period.
3. Women assigned to omega-3 fatty acid supplementation will report lower frequency and less VMS bother than women assigned to the placebo group at the end of a 12-week study period.

The omega-3 component of the study is double-blinded. For yoga, exercise, and usual activity, the outcomes assessors are blinded to the randomization assignments.

DETAILED DESCRIPTION:
Over 33 million U.S. women will transition through menopause in the next decade. Among women with natural menopause, the transition typically lasts four years, with a mean age at menopause of 51 years. Menstrual irregularity (90%) and vasomotor symptoms (VMS) (80%) are the most common symptoms associated with the transition. Hormone therapy has been the gold standard for treating VMS symptoms against which other therapies are measured. However, resistance to hormone therapy use due to its risks and side effects continues to fuel the search for safer alternatives.

This research study will evaluate three low risk interventions (yoga, exercise, and omega-3 supplements) compared to either a usual activity group or a placebo pill. This factorial design is motivated by the desire to have all women receive some intervention. Neither comparisons between yoga and exercise nor tests of interaction between the behavioral interventions (yoga, exercise, usual activity) and omega-3 motivated this design. However, these aspects can be examined in secondary analyses in a more rigorous fashion through this design than would be permitted by separate trials.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40-62 years.
* Menopausal, including:

  * Women who have had a bi-lateral oophorectomy;
  * Women with a uterus who have skipped 2 or more menstrual cycles with an amenorrhea interval of 60 or more days in the past 12 months;
  * Women without a uterus and who still have one or both ovaries, with FSH level greater than 20 mIU/mL and estradiol less than or equal to 50 pg/mL;
  * Women who are using the Mirena IUD or who have had an endometrial ablation and who still have one or both ovaries, with FSH level greater than 20 mIU/mL and estradiol less than or equal to 50 pg/mL.
* Having bothersome hot flashes and/or night sweats.
* In general good health as determined by medical history, blood pressure, and heart rate:

  * Absence of uncontrolled hypertension greater than 160/100;
  * Resting heart rate less than 110 beats per minute;.
  * No history of myocardial infarction, angina, or cerebrovascular events;.
  * No history of liver, renal disease, or uncontrolled seizure disorder.
  * Absence of uncontrolled metabolic disease (such as diabetes) and absence of current infectious disease (such as acute symptoms of mononucleosis) that would put staff and other participants at risk.
* Signed informed consent.

Exclusion Criteria:

* Use of hormone therapy or hormonal contraceptives (with the exception of the Mirena IUD) during the 2 months before enrollment. Vaginal postmenopausal estrogens allowed, with the exception of vaginal creams used more than 3 times a week.
* Use of any other therapy that is taken specifically for hot flashes, including prescription, over-the-counter, or herbal therapies, in the past month.
* Any current severe or unstable medical illness.
* Body mass index (BMI) of 37 or higher, based on measured height and weight.
* Severe uncorrected hearing or vision problems.
* Current, regular use of anti-coagulants 3 or more times per week, e.g. Coumadin, Heparin, Clopidogrel, aspirin at full dose (due to possible omega-3 supplement interaction).
* Drug or alcohol abuse in the past 1 year.
* Major severe depressive episode in the past 3 months.
* Diagnosis of psychosis or psychotic disorder.
* Pregnancy, intending pregnancy, or breastfeeding.
* Current participation in another drug trial or intervention study.
* Inability or unwillingness to complete the study procedures or interventions.
* Physical limitations that limit the ability to participate in yoga or exercise, for example:

  * Limited mobility (paralyzed, cannot walk 2 blocks);
  * Back problems (severe spine abnormality, sciatica, prior back surgery, spine fracture in the past 3 months);
  * musculoskeletal problems that limit the ability to walk on a treadmill or ride a stationary bicycle;
* Presence of any absolute contraindications to exercise testing and training, as defined by the American College of Sports Medicine.
* Practiced or attended any of the following in the prior 3 months:

  * Yoga, tai chi, qi gong, or meditation more than one time per week on average;
  * Aerobic exercise (more than 30 minutes a day on at least 3 days a week);
  * Inability to achieve 85% of heart rate reserve (HRR; the difference between maximum heart rate and resting heart rate) on graded exercise treadmill test.
* Severe allergy to soy (defined as life-threatening reaction to soy that would require medical intervention).
* Allergy or sensitivity to fish.
* Currently eating 4 or more servings of fish per week.
* Currently taking an omega-3 fish oil supplement more than twice per week in the past 4 weeks and unwilling to stop for 12 weeks. Interest women can stop all omega-3 supplements and reevaluate eligibility 4 weeks after stopping the omega-3 supplements.

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Frequency and bother of hot flashes measured by self-report diaries. | 12 weeks

SECONDARY OUTCOMES:
Frequency of hot flashes measured by objective biological marker. | 12 weeks
Anxiety, health- and menopause-related quality of life, depressed mood, and sleep (subjective by diaries and objective by sleep watch worn on wrist). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z. LaCroix, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Garnet Anderson, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Susan D Reed, MD, MPH, Principal Investigator — University of Washington/Group Health Research Institute; Katherine M Newton, PhD, Principal Investigator — Group Health Research Institute; Bette Caan, DrPH, Principal Investigator — Kaiser Permanente; Barbara Sternfeld, PhD, Principal Investigator — Kaiser Permanente; Janet Carpenter, PhD, RN, FAAN, Principal Investigator — Indiana University School of Medicine; Hadine Joffee, MD, MSc, Principal Investigator — Massachusetts General Hospital; Lee Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Kaiser Division of Research, Oakland, California
  - Indiana University, Indianapolis, Indiana
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- [Background] Sternfeld B, LaCroix A, Caan BJ, Dunn AL, Newton KM, Reed SD, Guthrie KA, Booth-LaForce C, Sherman KJ, Cohen L, Freeman MP, Carpenter JS, Hunt JR, Roberts M, Ensrud KE. Design and methods of a multi-site, multi-behavioral treatment trial for menopausal symptoms: the MsFLASH experience. Contemp Clin Trials. 2013 May;35(1):25-34. doi: 10.1016/j.cct.2013.02.009. Epub 2013 Feb 24. PMID 23462342
- [Derived] Diem SJ, LaCroix AZ, Reed SD, Larson JC, Newton KM, Ensrud KE, Woods NF, Guthrie KA. Effects of pharmacologic and nonpharmacologic interventions on menopause-related quality of life: a pooled analysis of individual participant data from four MsFLASH trials. Menopause. 2020 Oct;27(10):1126-1136. doi: 10.1097/GME.0000000000001597. PMID 32701665
- [Derived] Guthrie KA, Larson JC, Ensrud KE, Anderson GL, Carpenter JS, Freeman EW, Joffe H, LaCroix AZ, Manson JE, Morin CM, Newton KM, Otte J, Reed SD, McCurry SM. Effects of Pharmacologic and Nonpharmacologic Interventions on Insomnia Symptoms and Self-reported Sleep Quality in Women With Hot Flashes: A Pooled Analysis of Individual Participant Data From Four MsFLASH Trials. Sleep. 2018 Jan 1;41(1):zsx190. doi: 10.1093/sleep/zsx190. PMID 29165623
- [Derived] Jones SM, Guthrie KA, LaCroix AZ, Sternfeld B, Landis CA, Reed SD, Dunn A, Caan B, Cohen LS, Hunt J, Newton KM. Is heart rate variability associated with frequency and intensity of vasomotor symptoms among healthy perimenopausal and postmenopausal women? Clin Auton Res. 2016 Feb;26(1):7-13. doi: 10.1007/s10286-015-0322-x. Epub 2015 Dec 21. PMID 26691637
- [Derived] Guthrie KA, LaCroix AZ, Ensrud KE, Joffe H, Newton KM, Reed SD, Caan B, Carpenter JS, Cohen LS, Freeman EW, Larson JC, Manson JE, Rexrode K, Skaar TC, Sternfeld B, Anderson GL. Pooled Analysis of Six Pharmacologic and Nonpharmacologic Interventions for Vasomotor Symptoms. Obstet Gynecol. 2015 Aug;126(2):413-422. doi: 10.1097/AOG.0000000000000927. PMID 26241433
- [Derived] Newton KM, Reed SD, Guthrie KA, Sherman KJ, Booth-LaForce C, Caan B, Sternfeld B, Carpenter JS, Learman LA, Freeman EW, Cohen LS, Joffe H, Anderson GL, Larson JC, Hunt JR, Ensrud KE, LaCroix AZ. Efficacy of yoga for vasomotor symptoms: a randomized controlled trial. Menopause. 2014 Apr;21(4):339-46. doi: 10.1097/GME.0b013e31829e4baa. PMID 24045673
- [Derived] Cohen LS, Joffe H, Guthrie KA, Ensrud KE, Freeman M, Carpenter JS, Learman LA, Newton KM, Reed SD, Manson JE, Sternfeld B, Caan B, Freeman EW, LaCroix AZ, Tinker LF, Booth-Laforce C, Larson JC, Anderson GL. Efficacy of omega-3 for vasomotor symptoms treatment: a randomized controlled trial. Menopause. 2014 Apr;21(4):347-54. doi: 10.1097/GME.0b013e31829e40b8. PMID 23982113
- [Derived] Sternfeld B, Guthrie KA, Ensrud KE, LaCroix AZ, Larson JC, Dunn AL, Anderson GL, Seguin RA, Carpenter JS, Newton KM, Reed SD, Freeman EW, Cohen LS, Joffe H, Roberts M, Caan BJ. Efficacy of exercise for menopausal symptoms: a randomized controlled trial. Menopause. 2014 Apr;21(4):330-8. doi: 10.1097/GME.0b013e31829e4089. PMID 23899828
- [Derived] Newton KM, Carpenter JS, Guthrie KA, Anderson GL, Caan B, Cohen LS, Ensrud KE, Freeman EW, Joffe H, Sternfeld B, Reed SD, Sherman S, Sammel MD, Kroenke K, Larson JC, Lacroix AZ. Methods for the design of vasomotor symptom trials: the menopausal strategies: finding lasting answers to symptoms and health network. Menopause. 2014 Jan;21(1):45-58. doi: 10.1097/GME.0b013e31829337a4. PMID 23760428